CLINICAL TRIAL: NCT03141242
Title: Refining an Advance Care Planning Group Visit Intervention - A Novel Intervention to Engage Older Adults in Advance Care Planning.
Brief Title: ENgaging in Advance Care Planning Talks Group Visit Intervention
Acronym: ENACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1922
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Advance Care Planning; Primary Health Care
Keywords: Advance Care Planning; Group Medial Visit; Shared Medical Appointment

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENACT Group Visit (Active Comparator): Participants will engage in two 2-hour group visits related to advance care planning, including printed advance care planning resources.
  Interventions: Behavioral: ENACT group visit
- Mailed Resources (Placebo Comparator): Participants will receive printed advance care planning resources by mail.
  Interventions: Behavioral: Mailed Resources

INTERVENTIONS:
Behavioral: ENACT group visit — Participation in two 2 hour group visits about advance care planning.
  Arms: ENACT Group Visit
Behavioral: Mailed Resources — Participants will receive advance care planning resources in the mail with instructions to follow up with their primary care provider.
  Arms: Mailed Resources

SUMMARY:
The main goal of the ENACT (ENgaging in Advance Care planning Talks) Group Visit intervention is to integrate a patient-centered advance care planning process into primary care, ultimately helping patients to receive medical care that is aligned with their values. The ENACT Group Visit intervention involves two group discussions about advance care planning with 8-10 patients who meet for 2-hour sessions, one month apart, facilitated by a geriatrician and a social worker. This study will compare the ENACT Group Visit intervention to mailed advance care planning materials.

DETAILED DESCRIPTION:
This pilot feasibility randomized controlled study will determine the feasibility, acceptability and preliminary efficacy of the ENACT Group Visit intervention compared to a comparison arm.

The ENACT Group Visit intervention aims to engage patients in an interactive discussion of key ACP concepts and support patient-initiated ACP actions (i.e. choosing decision-maker(s), deciding on preferences during serious illness, discussing preferences with decision-makers and healthcare providers, and documenting advance directives). The group visits involve two 2-hour sessions, one month apart, facilitated by a geriatrician and a social worker. The ENACT Group Visit is based on an intervention manual that guides the structure, facilitator considerations, session format, and documentation and billing details. The discussions include sharing experiences related to ACP, considering values related to serious illness, choosing a surrogate decision-maker(s), flexibility in decision making, and having conversations with decision-makers and healthcare providers. The facilitators support an interactive discussion that promotes opportunities for patients to learn from others' experiences.

ELIGIBILITY:
Inclusion Criteria:

* 50 or older
* Receive primary care through UCHealth, Colorado, USA.

Exclusion Criteria:

* Severe cognitive impairment, known diagnoses of dementia
* Severe hearing loss or deafness

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Lum, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum HD, Jones J, Matlock DD, Glasgow RE, Lobo I, Levy CR, Schwartz RS, Sudore RL, Kutner JS. Advance Care Planning Meets Group Medical Visits: The Feasibility of Promoting Conversations. Ann Fam Med. 2016 Mar;14(2):125-32. doi: 10.1370/afm.1906. PMID 26951587
- [Derived] Lum HD, Dukes J, Daddato AE, Juarez-Colunga E, Shanbhag P, Kutner JS, Levy CR, Sudore RL. Effectiveness of Advance Care Planning Group Visits Among Older Adults in Primary Care. J Am Geriatr Soc. 2020 Oct;68(10):2382-2389. doi: 10.1111/jgs.16694. Epub 2020 Jul 29. PMID 32726475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ENACT Group Visit | Mailed Resources
Started | 55 | 55
Received Allocated Intervenion (Either attended group session or received mailed material, depending on arm) | 44 (11 subjects didn't attend their scheduled group session; all were included in ITT analysis) | 55
6 Month Interview | 51 | 49
Completed (Received 12 month Chart Review) | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ENACT Group Visit | Mailed Resources | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (5.3) | 77.2 (6.2) | 77.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 52 | 54 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 45 | 42 | 87
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 55 | 110
Relationship Status [Count of Participants; unit: Participants]
  Married/partnered | 34 | 35 | 69
  Widowed | 14 | 8 | 22
  Divorced or separated | 2 | 7 | 9
  Single | 5 | 5 | 10
Education Level [Count of Participants; unit: Participants]
  High school graduate | 3 | 5 | 8
  Some college | 9 | 17 | 26
  College graduate | 11 | 9 | 20
  Postgraduate or professional education | 32 | 24 | 56
Insurance Type [Count of Participants; unit: Participants]
  Medicare | 54 | 54 | 108
  Medicare Supplement | 28 | 33 | 61
  Medicaid | 0 | 2 | 2
  Tricare | 12 | 11 | 23
  Other | 11 | 8 | 19
Caregiver in the last 12 months [Count of Participants; unit: Participants]
  Yes | 12 | 12 | 24
  No | 43 | 43 | 86
Self-rated quality of life [Count of Participants; unit: Participants]
  Excellent | 22 | 22 | 44
  Fair | 6 | 7 | 13
  Good | 26 | 24 | 50
  Poor | 1 | 2 | 3
ACP documentation in EHR at baseline [Count of Participants; unit: Participants]
  Yes | 24 | 22 | 46
  No | 31 | 33 | 64
Self-report of memory concerns [Count of Participants; unit: Participants] | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Presence of Medical Decision-maker Documentation in the EHR
Description: An MDPOA form is in electronic medical chart or an orally appointed decision maker
Time Frame: 0, 6 months
Measure: Number; unit: participants
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 55 | 55
participants
  0 Months | 41 | 38
  6 Months | 51 | 40

2. Primary Outcome: Presence of Advance Directive in the EHR
Description: Presence of any advance directive document in the EHR (e.g., MDPOA, living will, Colorado MOST form)
Time Frame: 0 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 55 | 55
Participants
  Advance directive in EHR at 0 months | 24 | 22
  Advance directive in EHR at 6 months | 39 | 25

3. Secondary Outcome: Change in Advance Directive in Medical Record
Description: Any advance directive is present in the medical chart
Time Frame: 0, 3, 6, 12 months
Measure: Number; unit: participants
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 55 | 55
participants
  0 Months | 24 | 22
  3 Months | 38 | 24
  6 Months | 39 | 25
  12 Months | 42 | 28

4. Secondary Outcome: Change in Readiness to Engage in ACP (ACP Engagement Score)
Description: The Advance Care Planning (ACP) Engagement Scale will be used to assess readiness to engage in specific parts of the advance care planning process (i.e. signing official papers to name a medical decision maker; talking to the decision maker; talking to the doctor; signing official papers putting their wishes in writing). Items are rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate a higher level of engagement with the advance care planning behavior and a better outcome.
Time Frame: 0, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 51 | 49
units on a scale | 4.56 (.4) | 4.13 (.4)

5. Secondary Outcome: Change in Readiness to Chose a Surrogate Decision Maker
Description: Patient response to the question "How ready are you to sign official papers naming a medical decision maker to make medical decisions for you?". Responses were rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate more readiness and a better outcome.
Time Frame: 0, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 51 | 49
units on a scale
  0 months | 4.49 (0.9) | 4.25 (1.2)
  6 months | 4.8 (0.7) | 4.39 (1.0)

6. Secondary Outcome: Change in Readiness to Discuss Values and Care Preferences With Surrogate Decision Maker
Description: Patient response to the question "How ready are you to talk with your decision maker about what kind of medical care you would want if you were very sick or near the end of life?". Responses were rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate more readiness and a better outcome."
Time Frame: 0, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 51 | 49
units on a scale
  0 months | 4.65 (0.8) | 4.25 (1.1)
  6 months | 4.74 (0.8) | 4.28 (1.2)

7. Secondary Outcome: Readiness to Talk to Patient's Physician About Future Medical Care
Description: Patient response to the question "How ready are you to talk to your doctor about the kind of medical care you would want if you were very sick or near the end of life?". Responses were rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate more readiness and a better outcome.
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 55 | 55
units on a scale
  0 months | 3.47 (1.1) | 3.47 (1.3)
  6 months | 3.99 (1.2) | 3.59 (1.3)

8. Secondary Outcome: Readiness to Sign Official Papers About Medical Care
Description: Patient response to the question "How ready are you to sign official papers putting your wishes in writing about the kind of medical care you would want if you were very sick or near the end of life?". Responses were rated on a Likert scale, with possible scores ranging from 1-5. Higher scores indicate more readiness and a better outcome.
Time Frame: 0 and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 55 | 55
units on a scale
  0 months | 4.24 (1.0) | 4.04 (1.1)
  6 months | 4.69 (0.9) | 4.26 (1.1)

9. Other Pre Specified Outcome: Percent of Recruitment (Reach)
Description: Percent of individuals who participate of eligible patients, by clinic-based screening
Time Frame: From date of pre-screening until the date of participants' decision to enroll in study or not, up to 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Study Recruitment Rate: Participants will provide informed consent to participate in a randomized controlled trial of a two 2-hour group visit intervention related to advance care planning, including printed advance care planning resources (ENACT intervention arm) or a mailed advance care planning materials (mailed control arm)
Arm/Group | Study Recruitment Rate
Number analyzed (Participants) | 835
Participants | 110

10. Other Pre Specified Outcome: Percent of Retention
Description: Percent of individuals who complete the intervention and the 6 month follow up
Time Frame: Enrollment thru 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | ENACT Group Visit | Mailed Resources
Number analyzed (Participants) | 55 | 55
Participants | 51 | 49

ADVERSE EVENTS:
Time Frame: 6 months
Description: (Same as Clinical trials.gov) Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | ENACT Group Visit | Mailed Resources
All-Cause Mortality (participants affected / at risk) | 1/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 1/55 | 0/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENACT Group Visit (N=55) | Mailed Resources (N=55)
Psychological Distress (Psychiatric disorders) | 1 (1) | 0 (0) — Emotional triggering due to content of advance care planning and/or group visit discussion

LIMITATIONS AND CAVEATS:
20% (n=11) of participants randomized to the intervention arm did not attend a a group visit. They were included in intention to treat analysis, but this suggests feasibility and sustainability challenges and a need for pragmatic outreach and recruitment and flexible delivery options in practice. Possible selection bias in that there was a high baseline rate of ACP documentation. Low recruitment rate of 13% suggests need for more robust recruitment procedures for real-world implementation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03141242/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03141242/ICF_001.pdf